CLINICAL TRIAL: NCT00807521
Title: Reduction of the Cardiac Proapoptotic Stress Response by Dexamethasone in Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Steroid-induced Reduction of Surgical Stress Study
Acronym: STRESS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research question was integrated in other study protocol
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Christa Boer, Prof.dr. C. Boer, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 08/214
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Stenosis; Coronary Artery Bypass Graft Surgery
MeSH Terms: conditions — Coronary Stenosis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): High dose bolus of dexamethasone before surgery
  Interventions: Drug: Dexamethasone
- 2 (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Single high dose bolus of dexamethasone before surgery
  Arms: 1
Drug: Placebo — Placebo for dexamethasone
  Arms: 2

SUMMARY:
The stress response as induced by myocardial cellular damage during cardiac surgery may lead to myocardial stunning and apoptosis, and could therefore impair postoperative patient recovery. Surgical trauma typically induces the liberation of cytokines. Some of these cytokines are strongly associated with the initiation of intracellular proapoptotic pathways through activation of tyrosine kinases and integrins. The latter are known for their deteriorating effects on cardiac function and are strongly involved in cardiac remodeling. Dexamethasone is typically administered prior to cardiac surgery in order to especially reduce the release of proinflammatory cytokines. It has however never been investigated whether this additionally reduces proapoptotic signaling in the human heart, thereby eliminating risk factors for the induction of cardiac dysfunction. In the present study, the investigators therefore aim to investigate whether dexamethasone inhibits proapoptotic pathways in patients undergoing cardiac surgery. Furthermore, the investigators would like to elucidate whether this proposed effect of dexamethasone is related to the reduction of the stress response in the heart or indirectly by suppression of cytokine release. For this purpose the investigators will obtain cardiac biopsies and plasma from patients, who are randomly assigned to placebo or dexamethasone treatment and undergo on and off-pump coronary artery bypass grafting (CABG) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass surgery (CABG)
* Age 18-75 years
* Informed consent

Exclusion Criteria:

* Re-operations and emergency operations
* Patient with anemia (Hb < 5.0)
* Emergency operation
* Patients receiving blood transfusions < 3 months before operation
* Insulin depended diabetes mellitus
* Hepatic or renal failure
* Pregnancy
* Use of steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Expression of p38 in cultured cells and cardiac tissue | One week

SECONDARY OUTCOMES:
Pro-apoptotic signaling, precursor peptides of ANP (proANP), vasopressin (Copeptin), proET-1 and Adrenomedullin (proADM). Age, gender, length, body weight, hematocrit, Hb, leukocytes, surgery time, clamp time, CPB time | One week

CONTACTS AND LOCATIONS:
Overall Officials: Jan R. de Jong, MD, Principal Investigator — Amsterdam UMC, location VUmc; dr. Christa Boer, PhD, Study Chair — Amsterdam UMC, location VUmc; dr. Everaldo M. Redout, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- See also: General website of site — http://www.vumc.nl